CLINICAL TRIAL: NCT05897346
Title: Learning While Serving: Training Secondary School Students as Anti-smoke Ambassadors Using the Service-learning Model
Brief Title: Training Secondary School Students as Anti-smoke Ambassadors Using the Service-learning Model
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Katherine Lam, Research Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HP_Anti-smoke ambassadors
Record Dates: First submitted 2023-05-11; First posted 2023-06-09 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Smoking Cessation
Keywords: Adolescents; Training Activities; Knowledge, Attitudes, Practice; Self Efficacy
MeSH Terms: conditions — Smoking Cessation; Behavior

STUDY DESIGN:
Intervention Model Description: 14 clusters will be randomized to the intervention or control group using a 1:1 ratio by a research assistant using an independent computerized randomization sequence process.
Who Masked: Participant
Masking Description: The research assistant undertaking recruitment will be responsible for data collection and be blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Secondary school students will be required to join a 3-phase 'Learning while serving' program.
  Interventions: Other: 'Learning while serving' training program
- Control group (Other): Secondary school students will be only required to attend a 3-hour training workshops.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: 'Learning while serving' training program — The training program will involve training workshops, hands-on sessions, and a smoker referral competition.
  Arms: Intervention group
Other: Usual care — A 3-hour training workshops in the control group are regarded as usual care since the training workshops are also conducted regularly to other secondary or tertiary schools.
  Arms: Control group

SUMMARY:
Building the community's capacity by training youngsters to refer smokers to professional smoking cessation services offers a good strategy to support smoking cessation. Peer pressure is considered the most common reason for smoking in young people. Smoking cessation interventions that target peers are likely to have substantial effects. This health promotion project based on the service-learning model will provide opportunity for young people to learn and practice the AWARD model with hands-on experience under the supervision of nursing students who are considered experienced peer counselors.

DETAILED DESCRIPTION:
A hybrid type 1 effectiveness-implementation design will be adopted. A randomized sample of 368 students will be recruited from 14 secondary schools (Forms 2-4). The outcome measures will include demographic characteristics, the level of knowledge in smoking cessation and the AWARD model, the practice and attitude towards smoking cessation and the AWARD model, and the self-efficacy in using the AWARD model.

ELIGIBILITY:
Inclusion Criteria:

* secondary school students (Forms 2-4)

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The self-designed logbook for number of referrals at 6-month follow-up | at 6-month follow-up
  The number of smokers that referred to Youth Quitline will be recorded by using a self-designed logbook.

SECONDARY OUTCOMES:
The Knowledge towards Smoking Cessation and Tobacco Control Evaluation Questionnaire at baseline | at baseline
  Students' level of knowledge in smoking cessation and the AWARD model will be assessed by using the Knowledge towards Smoking Cessation and Tobacco Control Evaluation Questionnaire.
The Knowledge towards Smoking Cessation and Tobacco Control Evaluation Questionnaire at the end of training program | at the end of training program, an average of 2 years
  Students' level of knowledge in smoking cessation and the AWARD model will be assessed by using the Knowledge towards Smoking Cessation and Tobacco Control Evaluation Questionnaire.
The Knowledge towards Smoking Cessation and Tobacco Control Evaluation Questionnaire at 3-month follow-up | at 3-month follow-up
  Students' level of knowledge in smoking cessation and the AWARD model will be assessed by using the Knowledge towards Smoking Cessation and Tobacco Control Evaluation Questionnaire.
The Knowledge towards Smoking Cessation and Tobacco Control Evaluation Questionnaire at 6-month follow-up | at 6-month follow-up
  Students' level of knowledge in smoking cessation and the AWARD model will be assessed by using the Knowledge towards Smoking Cessation and Tobacco Control Evaluation Questionnaire.
The Knowledge towards Smoking Cessation and Tobacco Control Evaluation Questionnaire at 12-month follow-up | at 12-month follow-up
  Students' level of knowledge in smoking cessation and the AWARD model will be assessed by using the Knowledge towards Smoking Cessation and Tobacco Control Evaluation Questionnaire.
The Attitude/Practice towards Smoking Cessation and Tobacco Control Evaluation Questionnaire at baseline | at baseline
  Students' practice and attitude towards smoking cessation and the AWARD model will be assessed by using the Attitude/Practice towards Smoking Cessation and Tobacco Control Evaluation Questionnaire.
The Attitude/Practice towards Smoking Cessation and Tobacco Control Evaluation Questionnaire at the end of training program | at the end of training program, an average of 2 years
  Students' practice and attitude towards smoking cessation and the AWARD model will be assessed by using the Attitude/Practice towards Smoking Cessation and Tobacco Control Evaluation Questionnaire.
The Attitude/Practice towards Smoking Cessation and Tobacco Control Evaluation Questionnaire at 3-month follow-up | at 3-month follow-up
  Students' practice and attitude towards smoking cessation and the AWARD model will be assessed by using the Attitude/Practice towards Smoking Cessation and Tobacco Control Evaluation Questionnaire.
The Attitude/Practice towards Smoking Cessation and Tobacco Control Evaluation Questionnaire at 6-month follow-up | at 6-month follow-up
  Students' practice and attitude towards smoking cessation and the AWARD model will be assessed by using the Attitude/Practice towards Smoking Cessation and Tobacco Control Evaluation Questionnaire.
The Attitude/Practice towards Smoking Cessation and Tobacco Control Evaluation Questionnaire at 12-month follow-up | at 12-month follow-up
  Students' practice and attitude towards smoking cessation and the AWARD model will be assessed by using the Attitude/Practice towards Smoking Cessation and Tobacco Control Evaluation Questionnaire.
The Self-efficacy to Quit Evaluation Questionnaire at baseline | at baseline
  Students' self-efficacy in using the AWARD model will be measured by using the Self-efficacy to Quit Evaluation Questionnaire.
The Self-efficacy to Quit Evaluation Questionnaire at the end of training program | at the end of training program, an average of 2 years
  Students' self-efficacy in using the AWARD model will be measured by using the Self-efficacy to Quit Evaluation Questionnaire.
The Self-efficacy to Quit Evaluation Questionnaire at 3-month follow-up | at 3-month follow-up
  Students' self-efficacy in using the AWARD model will be measured by using the Self-efficacy to Quit Evaluation Questionnaire.
The Self-efficacy to Quit Evaluation Questionnaire at 6-month follow-up | at 6-month follow-up
  Students' self-efficacy in using the AWARD model will be measured by using the Self-efficacy to Quit Evaluation Questionnaire.
The Self-efficacy to Quit Evaluation Questionnaire at 12-month follow-up | at 12-month follow-up
  Students' self-efficacy in using the AWARD model will be measured by using the Self-efficacy to Quit Evaluation Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Wai Katherine Lam, Principal Investigator — School of Nursing, Hong Kong Polytechnic University
Locations (1):
- Katherine Lam, Hong Kong, Hong Kong,China, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lam KKW, Ho KY, Leung DYP, Wong AKC, Wu CST, Liu CQ, Mao T, Mak YW. Training secondary school students as anti-smoke ambassadors using the service-learning model: A cluster randomized controlled trial with hybrid type 1 effectiveness-implementation design study protocol. PLoS One. 2024 Nov 14;19(11):e0313404. doi: 10.1371/journal.pone.0313404. eCollection 2024. PMID 39541363